CLINICAL TRIAL: NCT03746366
Title: Imaging Beta-amyloid in Middle Age Alcoholics As a Mechanism That Increases Their Risk for Alzheimer's Disease
Brief Title: [C-11]PiB PET Imaging in Alcohol Use Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Rajesh Narendran, Professor of Radiology and Psychiatry, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO18080481; R01AA025247 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — 3-alpha-Hydroxysteroid Dehydrogenase (B-Specific); 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Intervention Model Description: [C-11]PiB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol use disorders (Experimental): [C-11]Pittsburgh Compound B (PiB) PET scan
  Interventions: Radiation: [C-11]; Drug: Pittsburgh Compound B
- Healthy controls (Experimental): [C-11]Pittsburgh Compound B (PiB) PET scan
  Interventions: Radiation: [C-11]; Drug: Pittsburgh Compound B

INTERVENTIONS:
Radiation: [C-11] — Radiolabel
Drug: Pittsburgh Compound B — Tracer

SUMMARY:
To determine whether alcoholics (AUD) have a greater rate of amyloid positivity (ABeta+) compared to an age-matched cognitively normal control group (HC).

DETAILED DESCRIPTION:
There is a long-established relationship between alcohol use disorders (AUD), cognitive impairments, and the development of dementia. Some, but not all basic data suggest that alcohol abuse can alter the expression of amyloid precursor protein, and the enzymes that process it. Thus, there is a need for in vivo PET studies to further investigate the relationship between AUD and AD and the mechanism through which alcohol abuse exerts its effect on this type of dementia. Here, we propose to use the amyloid Beta (ABeta) radiotracer carbon-11 labeled Pittsburgh Compound-B ([C-11]PiB) and PET (Klunk et al., 2004) to determine whether AUD increase the risk to be brain ABeta+ in middle aged adults.

ELIGIBILITY:
[A] Alcohol Use Disorder Subjects (AUD)

Inclusion Criteria:

1. Males or females between 40 and 65 years old
2. Fulfill DSM-5 criteria for alcohol use disorder of at least moderate severity
3. Current heavy drinking as defined in SAMHSA criteria (i.e., drinking 5 or more drinks on the same occasion on each of 5 or more days in the past 30 days)

Exclusion Criteria:

1. DSM-5 schizophrenia, schizoaffective disorder, bipolar disorder (SCID-5) and prior history of developmental disorders, such as Autism, Down's Syndrome, Intellectual disability.
2. A positive urine drug screen at screening for amphetamines, cocaine, methamphetamine, opioids, barbituates and PCP
3. History of severe unstable medical or neurological illnesses that could affect neuropsychological testing
4. History of cancer (other than skin or in situ prostate cancer) within the previous 5 years
5. Currently pregnant or breastfeeding
6. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year
7. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan
8. No first-degree relative with Alzheimer's disease or related dementias

(B) Healthy Control Subjects (HC)

Inclusion Criteria:

(1) Males or females between 40 and 65 years old

Exclusion criteria:

1. Current or past DSM-5 psychiatric and/or addictive disorders
2. Current heavy drinking as defined in SAMHSA criteria
3. History of severe unstable medical or neurological illnesses that could affect neuropsychological testing
4. History of cancer (other than skin or in situ prostate cancer) within the previous 5 years
5. Currently pregnant or breastfeeding
6. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year
7. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan
8. No first-degree relative with Alzheimer's disease or related dementias

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
[C-11]PIB + | Baseline
  positive/negative

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsbyurgh PET Facility, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flanigan MR, Royse SK, Cenkner DP, Kozinski KM, Stoughton CJ, Himes ML, Minhas DS, Lopresti B, Butters MA, Narendran R. Imaging beta-amyloid (Abeta) burden in the brains of middle-aged individuals with alcohol-use disorders: a [11C]PIB PET study. Transl Psychiatry. 2021 May 1;11(1):257. doi: 10.1038/s41398-021-01374-y. PMID 33934110